CLINICAL TRIAL: NCT03989960
Title: Application of Modified Intubation-surfactant-extubation (InSurE) Technique in Preterm Neonates With Respiratory Distress Syndrome
Brief Title: Modified Intubation-surfactant-extubation (InSurE) Technique in Preterm Neonates With Respiratory Distress Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOLISAN
Record Dates: First submitted 2019-06-17; First posted 2019-06-18 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Distress Syndrome of Newborn
Keywords: InSurE; LISA; SNIPPV
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LISA+SNIPPV group (Experimental): receives PS by the way of invasive surfactant administration technique and selects nasal synchronized intermittent positive pressure ventilation
  Interventions: Procedure: LISA+SNIPPV
- InSurE group (Active Comparator): receives intubation-surfactant- extubation technique and selects CPAP ventilation
  Interventions: Procedure: traditional InSurE

INTERVENTIONS:
Procedure: LISA+SNIPPV — The LISA+SNIPPV group receives PS by the way of invasive surfactant administration technique and selects nasal synchronized intermittent positive pressure ventilation.
  Arms: LISA+SNIPPV group
Procedure: traditional InSurE — The traditional InSurE group receives intubation-surfactant- extubation technique and selects CPAP ventilation.
  Arms: InSurE group

SUMMARY:
This study evaluates the less invasive surfactant administration (LISA) combined with synchronized nasal intermittent positive pressure ventilation (SNIPPV) technique in the treatment of respiratory distress syndrome (RDS) of preterm neonates. The modified InSurE group will receive "LISA + SNIPPV" technique, while the traditional InSurE group will receive the intubation, surfactant, extubation and CPAP technique.

ELIGIBILITY:
Inclusion Criteria:

1. premature infants with birth weight < 2500g and gestational age < 36+6 weeks;
2. High-risk premature infants with early symptoms of RDS or infants who are diagnosed clinically RDS.
3. the participating hospital obtained the consent of the Ethics Committee.
4. parental informed consents were obtained.

Exclusion Criteria:

1. severe congenital malformations.
2. severe cyanotic congenital heart disease (such as transposition of great artery, tetralogy of Fallot, etc.) which affects systemic hemodynamics.
3. congenital hereditary metabolic diseases.
4. parental informed consent was not obtained.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
the average duration of mechanical ventilation | 40 weeks
  the average duration of mechanical ventilation of each group
the duration of oxygen therapy | 40 weeks
  the duration of oxygen therapy of each group
the incidence of BPD | 28 days
  the incidence of BPD in each group

SECONDARY OUTCOMES:
Pulmonary Severity Score (PSC) | 1st, 2nd, 3rd, 7th, 14th, 28th days
  PSC was defined as FiO2 × support + medications, where FiO2 is the actual or 'effective' (for nasal cannula) FiO2; support is 2.5 for a ventilator, 1.5 for nasal continuous positive airway pressure, or 1.0 for nasal cannula or hood oxygen; and medications is 0.20 for systemic steroids for BPD, 0.10 each for regular diuretics or inhaled steroids, and 0.05 each for methylxanthines or intermittent diuretics. The scores can range from 0.21 to 2.95.
the incidence of complications | 40 weeks
  the incidence of complications (e.g. necrotizing enterocolitis, cholestasis, retinopathy of prematurity, extrauterine growth retardation)
oxygenation index and ventilation function (PaO2、a/APO2、FiO2、PaCO2) | the period of oxygen therapy
  oxygenation index and ventilation function (PaO2、a/APO2、FiO2、PaCO2)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqing Chen, Dr, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Plavka R, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GH, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2016 Update. Neonatology. 2017;111(2):107-125. doi: 10.1159/000448985. Epub 2016 Sep 21. PMID 27649091
- [Background] Patel RM, Kandefer S, Walsh MC, Bell EF, Carlo WA, Laptook AR, Sanchez PJ, Shankaran S, Van Meurs KP, Ball MB, Hale EC, Newman NS, Das A, Higgins RD, Stoll BJ; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Causes and timing of death in extremely premature infants from 2000 through 2011. N Engl J Med. 2015 Jan 22;372(4):331-40. doi: 10.1056/NEJMoa1403489. PMID 25607427
- [Background] Leone F, Trevisanuto D, Cavallin F, Parotto M, Zanardo V. Efficacy of INSURE during nasal CPAP in preterm infants with respiratory distress syndrome. Minerva Pediatr. 2013 Apr;65(2):187-92. PMID 23612264
- [Background] Sandri F, Plavka R, Ancora G, Simeoni U, Stranak Z, Martinelli S, Mosca F, Nona J, Thomson M, Verder H, Fabbri L, Halliday H; CURPAP Study Group. Prophylactic or early selective surfactant combined with nCPAP in very preterm infants. Pediatrics. 2010 Jun;125(6):e1402-9. doi: 10.1542/peds.2009-2131. Epub 2010 May 3. PMID 20439601
- [Background] Gopel W, Kribs A, Hartel C, Avenarius S, Teig N, Groneck P, Olbertz D, Roll C, Vochem M, Weller U, von der Wense A, Wieg C, Wintgens J, Preuss M, Ziegler A, Roth B, Herting E; German Neonatal Network (GNN). Less invasive surfactant administration is associated with improved pulmonary outcomes in spontaneously breathing preterm infants. Acta Paediatr. 2015 Mar;104(3):241-6. doi: 10.1111/apa.12883. PMID 25474712
- [Background] Kribs A, Hartel C, Kattner E, Vochem M, Kuster H, Moller J, Muller D, Segerer H, Wieg C, Gebauer C, Nikischin W, Wense Av, Herting E, Roth B, Gopel W. Surfactant without intubation in preterm infants with respiratory distress: first multi-center data. Klin Padiatr. 2010 Jan-Feb;222(1):13-7. doi: 10.1055/s-0029-1241867. Epub 2010 Jan 18. PMID 20084586
- [Background] Gopel W, Kribs A, Ziegler A, Laux R, Hoehn T, Wieg C, Siegel J, Avenarius S, von der Wense A, Vochem M, Groneck P, Weller U, Moller J, Hartel C, Haller S, Roth B, Herting E; German Neonatal Network. Avoidance of mechanical ventilation by surfactant treatment of spontaneously breathing preterm infants (AMV): an open-label, randomised, controlled trial. Lancet. 2011 Nov 5;378(9803):1627-34. doi: 10.1016/S0140-6736(11)60986-0. Epub 2011 Sep 29. PMID 21963186
- [Background] Niemarkt HJ, Hutten MC, Kramer BW. Surfactant for Respiratory Distress Syndrome: New Ideas on a Familiar Drug with Innovative Applications. Neonatology. 2017;111(4):408-414. doi: 10.1159/000458466. Epub 2017 May 25. PMID 28538236
- [Background] Kribs A, Roll C, Gopel W, Wieg C, Groneck P, Laux R, Teig N, Hoehn T, Bohm W, Welzing L, Vochem M, Hoppenz M, Buhrer C, Mehler K, Stutzer H, Franklin J, Stohr A, Herting E, Roth B; NINSAPP Trial Investigators. Nonintubated Surfactant Application vs Conventional Therapy in Extremely Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2015 Aug;169(8):723-30. doi: 10.1001/jamapediatrics.2015.0504. PMID 26053341
- [Background] Kanmaz HG, Erdeve O, Canpolat FE, Mutlu B, Dilmen U. Surfactant administration via thin catheter during spontaneous breathing: randomized controlled trial. Pediatrics. 2013 Feb;131(2):e502-9. doi: 10.1542/peds.2012-0603. Epub 2013 Jan 28. PMID 23359581
- [Background] More K, Sakhuja P, Shah PS. Minimally invasive surfactant administration in preterm infants: a meta-narrative review. JAMA Pediatr. 2014 Oct;168(10):901-8. doi: 10.1001/jamapediatrics.2014.1148. PMID 25089718
- [Background] Wu W, Shi Y, Li F, Wen Z, Liu H. Surfactant administration via a thin endotracheal catheter during spontaneous breathing in preterm infants. Pediatr Pulmonol. 2017 Jun;52(6):844-854. doi: 10.1002/ppul.23651. Epub 2017 Feb 2. PMID 28152280
- [Background] Klotz D, Porcaro U, Fleck T, Fuchs H. European perspective on less invasive surfactant administration-a survey. Eur J Pediatr. 2017 Feb;176(2):147-154. doi: 10.1007/s00431-016-2812-9. Epub 2016 Dec 9. PMID 27942865
- [Background] Heiring C, Jonsson B, Andersson S, Bjorklund LJ. Survey shows large differences between the Nordic countries in the use of less invasive surfactant administration. Acta Paediatr. 2017 Mar;106(3):382-386. doi: 10.1111/apa.13694. Epub 2017 Jan 4. PMID 27992064
- [Background] Aldana-Aguirre JC, Pinto M, Featherstone RM, Kumar M. Less invasive surfactant administration versus intubation for surfactant delivery in preterm infants with respiratory distress syndrome: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2017 Jan;102(1):F17-F23. doi: 10.1136/archdischild-2015-310299. Epub 2016 Nov 15. PMID 27852668
- [Background] Rigo V, Lefebvre C, Broux I. Surfactant instillation in spontaneously breathing preterm infants: a systematic review and meta-analysis. Eur J Pediatr. 2016 Dec;175(12):1933-1942. doi: 10.1007/s00431-016-2789-4. Epub 2016 Sep 27. PMID 27678511
- [Background] Keszler M, Sant'Anna G. Mechanical Ventilation and Bronchopulmonary Dysplasia. Clin Perinatol. 2015 Dec;42(4):781-96. doi: 10.1016/j.clp.2015.08.006. Epub 2015 Oct 1. PMID 26593078
- [Background] Jasani B, Nanavati R, Kabra N, Rajdeo S, Bhandari V. Comparison of non-synchronized nasal intermittent positive pressure ventilation versus nasal continuous positive airway pressure as post-extubation respiratory support in preterm infants with respiratory distress syndrome: a randomized controlled trial. J Matern Fetal Neonatal Med. 2016;29(10):1546-51. doi: 10.3109/14767058.2015.1059809. Epub 2015 Jul 28. PMID 26135774
- [Background] Ramos-Navarro C, Sanchez-Luna M, Sanz-Lopez E, Maderuelo-Rodriguez E, Zamora-Flores E. Effectiveness of Synchronized Noninvasive Ventilation to Prevent Intubation in Preterm Infants. AJP Rep. 2016 Jul;6(3):e264-71. doi: 10.1055/s-0036-1586205. PMID 27500013
- [Background] Moretti C, Gizzi C, Montecchia F, Barbara CS, Midulla F, Sanchez-Luna M, Papoff P. Synchronized Nasal Intermittent Positive Pressure Ventilation of the Newborn: Technical Issues and Clinical Results. Neonatology. 2016;109(4):359-65. doi: 10.1159/000444898. Epub 2016 Jun 3. PMID 27251453
- [Background] Lemyre B, Laughon M, Bose C, Davis PG. Early nasal intermittent positive pressure ventilation (NIPPV) versus early nasal continuous positive airway pressure (NCPAP) for preterm infants. Cochrane Database Syst Rev. 2016 Dec 15;12(12):CD005384. doi: 10.1002/14651858.CD005384.pub2. PMID 27976361
- [Background] Shi Y, Tang S, Zhao J, Shen J. A prospective, randomized, controlled study of NIPPV versus nCPAP in preterm and term infants with respiratory distress syndrome. Pediatr Pulmonol. 2014 Jul;49(7):673-8. doi: 10.1002/ppul.22883. Epub 2013 Sep 4. PMID 24039148
- [Background] Li W, Long C, Zhangxue H, Jinning Z, Shifang T, Juan M, Renjun L, Yuan S. Nasal intermittent positive pressure ventilation versus nasal continuous positive airway pressure for preterm infants with respiratory distress syndrome: a meta-analysis and up-date. Pediatr Pulmonol. 2015 Apr;50(4):402-9. doi: 10.1002/ppul.23130. Epub 2014 Nov 21. PMID 25418007
- [Background] Isayama T, Iwami H, McDonald S, Beyene J. Association of Noninvasive Ventilation Strategies With Mortality and Bronchopulmonary Dysplasia Among Preterm Infants: A Systematic Review and Meta-analysis. JAMA. 2016 Aug 9;316(6):611-24. doi: 10.1001/jama.2016.10708. PMID 27532916
- [Background] Owen LS, Manley BJ. Nasal intermittent positive pressure ventilation in preterm infants: Equipment, evidence, and synchronization. Semin Fetal Neonatal Med. 2016 Jun;21(3):146-53. doi: 10.1016/j.siny.2016.01.003. Epub 2016 Feb 26. PMID 26922562
- [Background] Lemyre B, Davis PG, De Paoli AG, Kirpalani H. Nasal intermittent positive pressure ventilation (NIPPV) versus nasal continuous positive airway pressure (NCPAP) for preterm neonates after extubation. Cochrane Database Syst Rev. 2017 Feb 1;2(2):CD003212. doi: 10.1002/14651858.CD003212.pub3. PMID 28146296
- [Background] Oncel MY, Arayici S, Uras N, Alyamac-Dizdar E, Sari FN, Karahan S, Canpolat FE, Oguz SS, Dilmen U. Nasal continuous positive airway pressure versus nasal intermittent positive-pressure ventilation within the minimally invasive surfactant therapy approach in preterm infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2016 Jul;101(4):F323-8. doi: 10.1136/archdischild-2015-308204. Epub 2015 Nov 9. PMID 26553376
- [Background] Gizzi C, Montecchia F, Panetta V, Castellano C, Mariani C, Campelli M, Papoff P, Moretti C, Agostino R. Is synchronised NIPPV more effective than NIPPV and NCPAP in treating apnoea of prematurity (AOP)? A randomised cross-over trial. Arch Dis Child Fetal Neonatal Ed. 2015 Jan;100(1):F17-23. doi: 10.1136/archdischild-2013-305892. Epub 2014 Oct 15. PMID 25318667
- [Background] Huang L, Mendler MR, Waitz M, Schmid M, Hassan MA, Hummler HD. Effects of Synchronization during Noninvasive Intermittent Mandatory Ventilation in Preterm Infants with Respiratory Distress Syndrome Immediately after Extubation. Neonatology. 2015;108(2):108-14. doi: 10.1159/000431074. Epub 2015 Jun 17. PMID 26107742